CLINICAL TRIAL: NCT01423448
Title: A Randomized Controlled Trial of an Online Bulletin Board for Depression
Brief Title: Effectiveness of an Online Bulletin Board for Depression: a Longitudinal Randomized Controlled Trial
Acronym: ShareIT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Recruitment of participants did not commence due to lack of available staff to run the trial.
Sponsor: Louise Farrer (Other)
Responsible Party: Sponsor-Investigator, Louise Farrer, Postdoctoral Research Fellow, Australian National University
Organization: Australian National University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CMHR-123; NHMRC Fellowship ref 525413 (Other Grant/Funding Number: National Health and Medical Research Council)
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Depression
Keywords: Depression; mental health; wellbeing; online bulletin board; online support group
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bulletin board (Experimental): Participants will be given access to the online bulletin board (intervention) for a 6 month period
  Interventions: Other: bulletin board
- Control (No Intervention): After 6 months participants allocated to the control group will receive access to the intervention

INTERVENTIONS:
Other: bulletin board — An asynchronous online bulletin board for people with experience of depression
  Arms: Bulletin board

SUMMARY:
This study is a randomised controlled trial that aims to examine the efficacy of an established online bulletin board for depression. It has been estimated that millions of people worldwide use peer-to-peer bulletin boards, forums or internet support groups (ISGs) for health conditions. However, little is known about the effectiveness of these groups in terms of symptom reduction or improvement in quality of life. The current project investigates the effectiveness of an established online bulletin board for depression available to the public. To our knowledge, this is the first randomised controlled trial of the effectiveness of a pre-existing, well-established online bulletin board for depression in the community. The aims of the project are to determine whether the bulletin board improves mental health, quality of life, and related outcomes among members of the community with high levels of self-reported psychological distress and previous history or current experience of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Internet access with email
3. Self-report of current or previous experience of depression

Exclusion Criteria:

1. Current participation in an online support group for depression
2. Diagnosis of bipolar disorder, schizophrenia, or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms: Centre for Epidemiological Studies - Depression Scale (CES-D) | Baseline
  20-item self -report measure of depression severity
Depressive symptoms: Centre for Epidemiological Studies - Depression Scale (CES-D) | 6 months post-baseline
  20-item self -report measure of depression severity
Depressive symptoms: Centre for Epidemiological Studies - Depression Scale (CES-D) | 12 months post-baseline
  20-item self -report measure of depression severity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Mental Health Research, The Australian National University, Canberra, Australian Capital Territory, Australia